CLINICAL TRIAL: NCT07166263
Title: Exploratory Study of NK510 Cell Therapy in the Treatment of Recurrent and Refractory Advanced Gastric Cancer and Colorectal Cancer
Brief Title: Safety and Efficacy of NK510 to Treat Gastric Cancer and Colorectal Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK510-13
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer (GC); Colorectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic therapy with NK510 via intravenous infusion (Experimental): Systemic therapy with NK510 via intravenous infusion combined with PD-L1 or other regimens selected by the investigator
  Interventions: Drug: NK510
- Intraperitoneal perfusion therapy with NK510 (Experimental): Intraperitoneal perfusion therapy with NK510 plus IL-2, PD-L1 or other regimens selected by the investigator for systemic therapy
  Interventions: Drug: NK510

INTERVENTIONS:
Drug: NK510 — NK510 will be administered through intravenous infusion, once a week for a total of six times.
  Arms: Systemic therapy with NK510 via intravenous infusion
Drug: NK510 — NK510 will be administered through intraperitoneal perfusion on D1, D4, and D7 of the first week for a total of 3 times, with each 3-week cycle constituting a total of 2 cycles.
  Arms: Intraperitoneal perfusion therapy with NK510

SUMMARY:
This study will evaluate the safety and efficacy of NK510 in the treatment of relapsed and refractory advanced gastric cancer and colorectal cancer.NK510 will be administered by intravenous infusion for systemic therapy and intraperitoneal perfusion therapy. The safety and efficacy of this treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, regardless of gender.
2. Gastric cancer and colorectal cancer that are inoperable and unresectable with radiotherapy: For gastric cancer, molecular diagnosis confirms that it is not AFP-producing gastric cancer.
3. Progressive disease or recurrence after receiving ≥ 2 lines of treatment.
4. Patients are divided into two groups (Group A and Group B) based on the presence or absence of peritoneal metastasis. The criteria for determining peritoneal metastasis are as follows:

   1. Drained ascites ≥ 500ml, or B-ultrasound/CT in the supine position shows ascites depth ≥ 3cm.
   2. Peritoneal metastasis confirmed by any of the following criteria:

   i. Positive for exfoliated cancer cells in ascites. ii. Diagnosed as peritoneal metastatic carcinoma by imaging and symptoms. iii. Peritoneal metastasis confirmed by abdominal exploration. iv. Ascites confirmed as exudate by routine ascites examination and ascites biochemistry.
5. At least one measurable lesion on CT or MRI according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors).
6. ECOG performance status of 0-2.
7. Expected survival period ≥ 3 months.
8. Able to comply with the study protocol and follow-up procedures, and voluntarily sign the informed consent form for participation in this study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects with central nervous system (CNS) metastases and/or carcinomatous meningitis with obvious symptoms.
3. A history of other malignant tumors within the past 3 years.
4. Subjects with active, known or suspected autoimmune diseases [excluding type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, or alopecia), or diseases that are not expected to relapse without external triggers].
5. Subjects with a history of immunodeficiency, including positive HIV test results, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
6. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities such as ventricular arrhythmias requiring clinical intervention, third-degree atrioventricular block, etc.; QTc interval > 480 ms on 12-lead electrocardiogram at rest; acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events within 6 months before enrollment; New York Heart Association (NYHA) cardiac function classification ≥ class II or left ventricular ejection fraction (LVEF) < 50%; clinically uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | 6 weeks
  To evaluate the DLT during N510 treatment
Overall response rate (ORR) | 6 weeks
  Effectiveness Metrics
Puncture-free survival (PuFS) | 6 weeks
  Effectiveness Metrics

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Affiliated to the Medical School of Nanjing University, Nanjing, Jiangsu, China